CLINICAL TRIAL: NCT00218686
Title: Supplement to the Long-term Impact of a Network Outreach Intervention
Brief Title: A Network Intervention for Prevention of HIV Infection in Chennai, India - 1
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: In ability to obtain Indian governmental approval from the study from NACO
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DESPR DA013142; R01-13142-1; NIDA-13142-1
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: HIV; injection drug use; social networks
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): behavioral social network risk reduction intervention
  Interventions: Behavioral: psychoeducational
- 2 (Active Comparator): voluntary counseling and testing (VCT
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: psychoeducational — psychoeducational
  Arms: 1
Behavioral: control — VTC
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate a peer-based HIV prevention intervention that targets active injection drug users and their drug and sex partners in Chennai India.

DETAILED DESCRIPTION:
The intervention to be tested in this study draws upon theoretical and empirical evidence suggesting that peer educator programs can have significant effects on the risk-related behaviors of both the educators and the peers whom they educate. Specifically, through group and individual focused sessions, participants learn and practice skills designed to reduce drug and sex related risk behaviors. Furthermore, individuals and their main risk partners attend a training session that focuses on risk reduction within their relationship.

ELIGIBILITY:
Inclusion Criteria:

* drug users
* network members

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
needle sharing | 3 month
condom use | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carl Latkin, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- YRG Care, Chennai, Tamil Nadu, India